CLINICAL TRIAL: NCT04606004
Title: Perianal Maceration in Pediatric Ostomy Closure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Robert Morris University (Unknown)
Responsible Party: Principal Investigator, Victoria Morando, Registered Nurse, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY20030192
Record Dates: First submitted 2020-10-21; First posted 2020-10-28 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Perianal Dermatitis; Diaper Dermatitis; Postoperative Complications; Colostomy Site; Ileostomy - Stoma
MeSH Terms: conditions — Diaper Rash; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (standard of care + stool application) (Experimental): In addition to standard of care, they will apply stool from the stoma bag 4 weeks prior, twice daily for 10 minutes at a time.
  Interventions: Other: Stool application; Other: Standard of care skincare
- Control group (standard of care) (Active Comparator): Will follow standard of care for skin care pre-operatively. They will not be applying ostomy stool output to the skin but can apply an OTC skin barrier such as Aquaphor, Desitin, or Vitamin A&D if the patient is experiencing skin redness from urine incontinence.
  Interventions: Other: Standard of care skincare

INTERVENTIONS:
Other: Stool application — Application of stool from the stoma bag 4 weeks prior, twice daily for 10 minutes at a time. However, with the stool application no barrier cream will be applied to the skin in order for the stool to achieve penetrance to the skin. Stool application will include removing any barrier creams gently, applying a thin layer of stool with a surface area shown in illustration to ensure consistent coverage, and placing a diaper on the subject. Depending on the type of the participant's ostomy, a medication cup, syringe, and/or tongue blade provided by the researchers, may be used to aid in the application of stool. After 10 minutes of application, the caregiver or inpatient healthcare provider will remove the entire thin layer of stool gently without excessive friction, just enough to remove the stool, a dabbing motion is preferred.
  Arms: Experimental (standard of care + stool application)
Other: Standard of care skincare — Standard of care for skin care pre-operatively: which is either no application of barrier cream, or an application of an over the counter (OTC) skin barrier such as Aquaphor, Desitin, or Vitamin A&D if the patient is experiencing skin redness from urine incontinence.
  Standard of care skin creams post op: 3M no-sting immediately post op, once begin stooling- stoma powder, 3M no-sting, Critic-aid thick barrier paste will be applied to the skin.

SUMMARY:
This pilot study will explore whether preoperative application of stool from the stoma bag to the perianal area will prevent/ decrease postoperative perianal maceration in pediatric ostomy closure patients. It will also explore the overall safety and feasibility of this pilot study for larger randomized control trials. There will be a control group and an intervention group. The intervention group will apply stool from the stoma bag approximately 4 weeks prior to ostomy closure and fill out a compliance log and upload pictures weekly to the MyCHP (My Children's Hospital) portal. A validated diaper dermatitis score will be utilized in this study.

DETAILED DESCRIPTION:
After consent, participants will be assigned to either a treatment group or control group using a 2-group comparative pilot design. For this pilot study to ensure adequate balance, subjects will be assigned using every other technique. After consent is obtained, a one-time pH stool sample will be collected either at the outpatient visit or at the inpatient's bedside.

Pre-Operatively (about 4 weeks prior to ostomy closure)

Intervention Group:

The parent or the inpatient healthcare provider (if patient is hospitalized at any point within the 4 weeks prior to ostomy closure) will follow standard of care for skin care pre-operatively, which is either no application of barrier cream, or an application of an over the counter skin barrier such as Aquaphor, Desitin, or Vitamin A&D if the patient is experiencing skin redness from urine incontinence. In addition to standard of care, they will apply stool from the stoma bag 4 weeks prior, twice daily for 10 minutes at a time. However, with the stool application no barrier cream will be applied to the skin in order for the stool to achieve penetrance to the skin. After 10 minutes of application, the caregiver or inpatient healthcare provider will remove the entire thin layer of stool gently without excessive friction, just enough to remove the stool, a dabbing motion is preferred. Parents will be asked to upload images of their child's diaper area at least once weekly onto the MyCHP Portal (if their child is not inpatient) in order to monitor their skin for breakdown from and while performing the intervention. If at any time redness occurs, the parent will be asked to upload an additional picture to the MyCHP Patient Portal for investigator/clinician review or for visual inspection (if inpatient) and corresponding measurement of perianal skin breakdown. Upon visual inspection or image inspection, the co-investigator/ clinician will provide review, corresponding measurement with a validated diaper dermatitis scale, and provide appropriate clinical guidance.

Compliance and Assessment: A preoperative compliance log will be used with every stool application by the parent at home or healthcare provider. This log will ask who applied the stool, how long stool was on the skin, description of stool, skin description, what brand of diapers and wipes were used, diet information, etc. They will notify the researchers if there are worsening skin concerns at home. Weekly and as needed images of buttocks areas will be uploaded into the CHP Patient Portal for clinical/research review by the parent, or weekly visual inspections as needed assessments by the principal investigator or co-investigators for hospitalized patients pre-operatively. On day of closure there will be a one time assessment to get a baseline assessment of skin prior to surgery. Compliance logs will also be turned in at this time.

Control Group:

Skin care inpatient and outpatient:

Will follow standard of care for skin care pre-operatively. They will not be applying ostomy stool output to the skin but can apply an over the counter skin barrier such as Aquaphor, Desitin, or Vitamin A&D if the patient is experiencing skin redness from urine incontinence. One-time assessment on day of closure to ensure no application of stool to buttocks area was conducted during pre-operative period and to get a baseline assessment.

------ Post Operatively Post op day 1 - 1st post-operative appt (approximately 1-month) Intervention Group and Control Group

Standard of care skin creams including 3M no-sting immediately post op, once begin stooling- stoma powder, 3M no-sting, Critic-aid thick barrier paste will be applied to the skin. The parents and/or health care providers will use home-made wipes (water moistened gauze) to clean the skin. Healthcare providers and/or parents will provide q2h diaper checks. If there is worsening of the skin condition or concerns, the healthcare provider will notify the enterostomal nurse and place a new skin care consult. Additional interventions suggested by the enterostomal nurse may include BID(twice daily) Aveeno soaks, BID Domeboro soaks, or blow by 02 to the buttocks.

With each diaper change, the caregiver and/or the nurse will assess the child's diaper area.

* Twice weekly and as needed images of buttocks areas will be uploaded onto the CHP (Children's Hospital of Pittsburgh) Patient Portal for both groups once outpatient. The investigators will provide review and corresponding measurement with a validated diaper dermatitis scale.
* Weekly and as needed visual inspections of buttocks area for clinical/research review when still inpatient.

At postoperative visit:

Return of preoperative log if previously forgot. The parent will fill out a questionnaire at this time. There will be one more assessment of their skin at this appointment.

Electronic Medical Record (EMR) Review An electronic medical record review will be performed to collect information necessary for this study including demographic data (age, gender, race), gestational age, initial diagnosis, comorbidities, type of ostomy, duration of ostomy, reason for stoma closure, height/weight percentiles (at birth & at closure), formula vs breast milk, diet at time of closure, diet information, inpatient vs outpatient, intervention vs control, length of stay, medication use (antibiotics, cholestyramine, Imodium, Metamucil, etc.), post-operative complications, skin assessments, any additional skin care interventions (aveeno soaks, domeboro soaks, blow by 02, nystatin, etc.), labs, length of stay, previous ostomy complications/revisions/surgeries, and if discharged home prior to closure,etc.

Compliance log Compliance logs will be reviewed for the following: If they were compliant/non-compliant with the study, type of diapers (brand, cloth, pull-ups), type of water used to clean (fresh vs well), frequency of feeds, diet, etc.

ELIGIBILITY:
Inclusion Criteria:

* Ostomy closure (colostomy & ileostomy)
* ages 3 years & under (still in diapers)
* male & female
* Scheduled ostomy closure in approximately 4 weeks.
* The legal guardian/parent of subject must have a personal device, such as a cell phone, that has access to internet in order to sign on to the MyCHP Portal.
* Participants must be enrolled in the MyCHP Portal.

Exclusion Criteria:

* Patients with a history of hypersensitive skin
* dermatological diagnosis
* ostomies other than colostomies/ileostomies
* ages older than 3 years
* Subjects who are not enrolled in the MyCHP Portal.
* Subjects with parents who do not have a personal device, such as a cell phone, or access to internet.

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Perianal skin maceration in the group receiving the intervention vs. the control group | from enrollment to the follow up postoperative appointment (approximately 4 weeks after surgery)
  this will be measured by uploading pictures or visual inspections and utilizing a validated diaper dermatitis scale (total severity score for the scale is 0-6, a higher score (6) indicates a worse outcome)

SECONDARY OUTCOMES:
The number & identification of influencing characteristics/variables of perianal skin breakdown | from enrollment to the follow up postoperative appointment (approximately 4 weeks after surgery)
  This will be done by doing a retrospective chart review and by reviewing the compliance log and parent questionnaire. The compliance log & parent questionnaire will be asking diaper brand, diet, stool consistency, etc. This will be determined by statistical analysis and by looking at diaper dermatitis scores via the validated scale (total severity score for the scale is 0-6, a higher score (6) indicates a worse outcome)
Incidence of complications (safety and tolerability of intervention) from application of stool between ileostomies vs. colostomies | from enrollment to the follow up postoperative appointment (approximately 4 weeks after surgery)
  this will be measured by uploading pictures or visual inspections and utilizing a validated diaper dermatitis scale (total severity score for the scale is 0-6, a higher score (6) indicates a worse outcome)
Explore parent compliance of application of stool at home vs. staff (RN) compliance of application of stool when inpatient | from enrollment to the follow up postoperative appointment (approximately 4 weeks after surgery)
  This will be done by reviewing the preoperative compliance log. The compliance log has a section to record when the application was performed and by who. (Should be twice daily 4 weeks prior to ostomy closure).

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Morando, RN, Principal Investigator — University of Pittsburgh; Kelly Austin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: Approximately 6- 9months following publication. No end date.
Access Criteria: Individual participant data that underlie the results reported in this article, after deidentification. With whomever would like to access it for any purpose. Mechanism yet to be determined.

REFERENCES:
- [Background] Dasgupta R, Langer JC. Evaluation and management of persistent problems after surgery for Hirschsprung disease in a child. J Pediatr Gastroenterol Nutr. 2008 Jan;46(1):13-9. doi: 10.1097/01.mpg.0000304448.69305.28. PMID 18162828
- [Background] Gray M. Incontinence-related skin damage: essential knowledge. Ostomy Wound Manage. 2007 Dec;53(12):28-32. PMID 18184980
- [Background] Heimall LM, Storey B, Stellar JJ, Davis KF. Beginning at the bottom: evidence-based care of diaper dermatitis. MCN Am J Matern Child Nurs. 2012 Jan-Feb;37(1):10-6. doi: 10.1097/NMC.0b013e31823850ea. PMID 22072018
- [Background] Keller DS, Khorgami Z, Swendseid B, Khan S, Delaney CP. Identifying causes for high readmission rates after stoma reversal. Surg Endosc. 2014 Apr;28(4):1263-8. doi: 10.1007/s00464-013-3320-x. Epub 2013 Nov 27. PMID 24281432
- [Background] Babuna Kobaner G, Sun GP, Ozkaya E. A recalcitrant case of Jacquet erosive diaper dermatitis after surgery for Hirschsprung disease in a boy with Waardenburg-Shah syndrome. Dermatol Online J. 2018 Jun 15;24(6):13030/qt8fk4t4rm. PMID 30142718
- [Background] Lim YSL, Carville K. Prevention and Management of Incontinence-Associated Dermatitis in the Pediatric Population: An Integrative Review. J Wound Ostomy Continence Nurs. 2019 Jan/Feb;46(1):30-37. doi: 10.1097/WON.0000000000000490. PMID 30608338
- [Background] Rodriguez-Poblador J, Gonzalez-Castro U, Herranz-Martinez S, Luelmo-Aguilar J. Jacquet erosive diaper dermatitis after surgery for Hirschsprung disease. Pediatr Dermatol. 1998 Jan-Feb;15(1):46-7. doi: 10.1046/j.1525-1470.1998.1998015046.x. PMID 9496804
- [Background] Shin HT. Diaper dermatitis that does not quit. Dermatol Ther. 2005 Mar-Apr;18(2):124-35. doi: 10.1111/j.1529-8019.2005.05013.x. PMID 15953142
- [Background] Tamaki K, Yokomori K. Diaper dermatitis with granuloma following surgery for Hirschsprung's disease. J Dermatol. 1987 Jun;14(3):262-5. doi: 10.1111/j.1346-8138.1987.tb03573.x. No abstract available. PMID 3312348
- See also: Skin benefits from continuous topical administration of a zinc oxide/petrolatum formulation by a novel disposable diaper. — https://www.ncbi.nlm.nih.gov/pubmed/11720074
- See also: Effects of potato-derived protease inhibitors on perianal dermatitis after colon resection for long-segment hirschsprung's disease. — https://www.ncbi.nlm.nih.gov/pubmed/22573429
- See also: Prevention of diaper dermatitis in infants-a literature review. — https://www.ncbi.nlm.nih.gov/pubmed/24890321
- See also: Etiologic factors in diaper dermatitis: the role of feces. — https://www.ncbi.nlm.nih.gov/pubmed/3513143
- See also: Faecal composition after surgery for hirschsprung's disease — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC1546124/
- See also: Factors determining the severity of perianal dermatitis after enterostoma closure of pediatric patients — http://resolver.ebscohost.com/openurl?sid=OVID%3amedline&pmid=15689222&issn=0011-9059&isbn=&volume=44&issue=2&spage=168&date=2005&title=International+Journal+of+Dermatology&atitle=Factors+determining+the+severity+of+perianal+dermatitis+after+enterostoma+closure+of+pediatric+patients.&aulast=Tokar&site=ftf-live